CLINICAL TRIAL: NCT04416984
Title: A Single-Arm, Open-Label, Phase 1/2 Study Evaluating the Safety, Efficacy, and Cellular Kinetics/Pharmacodynamics of ALLO-501A, an Anti-CD19 Allogeneic CAR T Cell Therapy, and ALLO-647, an Anti-CD52 Monoclonal Antibody, in Subjects with Relapsed/Refractory Large B-Cell Lymphoma (LBCL)
Brief Title: Safety and Efficacy of ALLO-501A Anti-CD19 Allogeneic CAR T Cells in Adults with Relapsed/Refractory Large B Cell Lymphoma, Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma (ALPHA2)
Acronym: ALPHA2
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Allogene Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALLO-501A-201
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Relapsed or Refractory Large B Cell Lymphoma, Relapsed or Refractory Chronic Lymphocytic Leukemia, Relapsed or Refractory Small Lymphocytic Lymphoma
Keywords: CAR T; Cell Therapy; Allogeneic Cell Therapy; Cellular Immuno-therapy; AlloCAR T; ALLO-501A; ALLO-647; LBCL; Lymphoma; Large B-Cell Lymphoma; Cema-cel; Cemacabtagene ansegedleucel; Leukemia; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL
MeSH Terms: conditions — Recurrence; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ALLO-501A, ALLO-647 (Experimental)
  Interventions: Genetic: ALLO-501A; Biological: ALLO-647; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Genetic: ALLO-501A — ALLO-501A is an allogeneic CAR T cell therapy targeting CD19
Biological: ALLO-647 — ALLO-647 is a monoclonal antibody that recognizes a CD52 antigen
Drug: Fludarabine — Chemotherapy for lymphodepletion
Drug: Cyclophosphamide — Chemotherapy for lymphodepletion

SUMMARY:
This is a single-arm, open label, multicenter Phase 1/2 study evaluating ALLO-501A in adult subjects with R/R LBCL and CLL/SLL. The purpose of the ALPHA2 study is to assess the safety, efficacy, and cell kinetics of ALLO-501A in adults with relapsed or refractory large B-cell lymphoma and assess the safety of ALLO-501A in adults with relapsed or refractory chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) after a lymphodepletion regimen comprising fludarabine, cyclophosphamide, and ALLO-647.

ELIGIBILITY:
Inclusion Criteria:

For subjects with LBCL:

* Histologically confirmed diagnosis of relapsed/refractory large B-cell lymphoma at last relapse per WHO 2017
* At least 1 measurable lesion at time of enrollment
* Relapsed or refractory disease after at least 2 lines of chemotherapy
* Absence of significant donor (product)-specific anti-HLA antibodies (DSA) at screening (Note: Only applicable for Phase 2)

For subjects with CLL/SLL:

* Diagnosis of CLL/SLL
* Relapsed/refractory disease
* Subjects relapsed/refractory to BTKi therapy and high-risk disease
* Subjects relapsed/refractory with 2 or more lines of therapy including BTKi and BCL-2 inhibitor (venetoclax)
* At least 1 measurable lesion at time of enrollment

For all subjects:

* Male or female subjects ≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
* Adequate hematological, renal, and liver function

Exclusion Criteria:

* Active central nervous system (CNS) involvement by malignancy
* Current thyroid disorder (including hyperthyroidism), except for subjects with hypothyroidism controlled on a stable dose of hormone replacement therapy
* Any other active malignancies that required systemic treatment within 3 years prior to enrollment
* Radiation therapy within 2 weeks prior to ALLO-647
* Prior irradiation to >25% of the bone marrow
* Hypocellular bone marrow for age by institutional standard as determined from a bone marrow biopsy performed at time of screening (Note: Only applicable for Phase 2).
* Autologous hematopoietic stem cell transplant (HSCT) within last 6 months (24 weeks)
* Systemic anti-cancer therapy within 2 weeks prior to receiving ALLO-647

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Proportion of subjects experiencing Dose Limiting Toxicities (DLT) at increasing doses of ALLO-501A | 28 days
  Dose limiting toxicity is defined as protocol-defined ALLO-501A-related adverse events with onset within 28 days following infusion
Phase 1a: Proportion of subjects experiencing Dose Limiting Toxicity with ALLO-647 in combination with fludarabine/cyclophosphamide administered prior to ALLO-501A | 33 days
  DLT is defined as protocol-defined ALLO-647-related adverse events with onset within 33 days following 1st infusion
Phase 1b: Frequency and severity of ALLO-501A treatment-emergent adverse events (AEs), serious AEs, and AEs of special interest | Up to 60 months
Phase 2: Overall Response Rate (ORR) assessed per Independent Review Committee (IRC) | Up to 60 months
  ORR defined as assessment of CR and PR using Lugano classification criteria 2014

SECONDARY OUTCOMES:
Phase 1a, 1b, and 2: Duration of Response (DOR) assessed per IRC (Phase 2 only) and per investigator | Up to 60 months
  DOR is defined only for subjects who experience an objective response and is the time from the first objective response to disease progression or death, whichever comes first per (Cheson et al, 2014)
Phase 1a, 1b, and 2: Overall Response Rate (ORR) assessed per investigator | Up to 60 months
Phase 1a, 1b, and 2: Best overall response (CR, PR, SD, PD) assessed per IRC (Phase 2 only) and per investigator | Up to 60 months
  CR Complete Response, PR Partial Response, SD Stable Disease, PD Progressive Disease
Phase 1a, 1b, and 2: Progression Free Survival (PFS) assessed per IRC (Phase 2 only) and per investigator | Up to 60 months
  PFS, defined as time from the enrollment date to progression, relapse, or death
Phase 1a, 1b, and 2: Time to Response (TTR) assessed per IRC (Phase 2 only) and per investigator | Up to 60 months
  TTR, defined as the time from the enrollment date to the first observed response
Phase 1a, 1b, and 2: Overall Survival (OS) | Up to 60 months
  OS, defined as the time from the enrollment date to death
Phase 1a, 1b, and 2: Depth of lymphodepletion as assessed by lymphocyte count | Up to 9 months
Phase 1a, 1b, and 2: Duration of lymphodepletion as assessed by lymphocyte recovery | Up to 9 months
Phase 1a, 1b, and 2: Serum concentration of ALLO-647 as measured by microgram per microliter for use in a population PK model | Up to 9 months
Phase 1a, 1b, and 2: ALLO-501A expansion assessed by peak blood concentration (Cmax) | Up to 9 months
Phase 1a, 1b, and 2: ALLO-501A expansion assessed by area under the curve (AUC) | Up to 9 months
Phase 1a, 1b, and 2: ALLO-501A persistence assessed by peak blood concentration (Cmax) | Up to 9 months
Phase 1a, 1b, and 2: ALLO-501A persistence assessed by area under the curve (AUC) | Up to 9 months
Phase 1a, 1b, and 2: Pharmacodynamics will be evaluated on host T cell counts | Up to 9 months
Phase 1a, 1b, and 2: The incidence of anti-drug antibodies against ALLO-501A scFv and/or TALEN® | Up to 9 months
Phase 1a, 1b, and 2: The incidence of anti-drug antibodies against ALLO-647 | Up to 9 months
Phase 1a, 1b, and 2: Adverse Events (AEs) as characterized by preferred term, frequency, severity timing, seriousness, and relationship to ALLO-501A | Up to 60 months
  The incidence and severity of Cytokine Release Syndrome (CRS), Graft-Versus-Host Disease (GVHD), infections, cytopenias, and neurotoxicity
Phase 1a, 1b, and 2: AEs as characterized by preferred term, frequency, severity, timing, seriousness, and relationship to ALLO-647 | Up to 60 months
  The incidence of infusion-related reactions, cytopenias, and infections
Phase 1a, 1b, and 2: The incidence and severity of clinically significant laboratory toxicities and relationship to ALLO-647 | Up to 60 months

CONTACTS AND LOCATIONS:
Locations (23):
- United States (18):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - City of Hope, Duarte, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford Cancer Institute, Palo Alto, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami, Miami, Florida
  - Advent Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital - Atlanta, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Norton Cancer Institute, Louisville, Kentucky
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt Ingram Cancer Center, Nashville, Tennessee
  - St. David's South Austin Medical Center, Austin, Texas
  - Texas Oncology, Dallas, Texas
  - MD Anderson Cancer Center - University of Texas, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
- Canada (2):
  - QEII Health Sciences Centre-VG Site, Halifax, Nova Scotia
  - CHU de Québec -Université Laval; Hôpital de l'Enfant-Jésus, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Locke FL, Munoz JL, Tees MT, Lekakis LJ, de Vos S, Nath R, Stevens DA, Malik SA, Shouse GP, Hamadani M, Oluwole OO, Perales MA, Miklos DB, Fisher PW, Feng A, Navale L, Le Gall JB, Neelapu SS. Allogeneic Chimeric Antigen Receptor T-Cell Products Cemacabtagene Ansegedleucel/ALLO-501 in Relapsed/Refractory Large B-Cell Lymphoma: Phase I Experience From the ALPHA2/ALPHA Clinical Studies. J Clin Oncol. 2025 May 10;43(14):1695-1705. doi: 10.1200/JCO-24-01933. Epub 2025 Feb 13. PMID 39946666